CLINICAL TRIAL: NCT07175909
Title: Proteomics Analysis of Human Tears in the Diagnosis and Management of Dry Eye Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSE Sung Hei Jimmy, Assistant Professor of Practice, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: HSEARS20210311002
Record Dates: First submitted 2025-09-06; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye Disease (DED); Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DED Treatment Arm (Active Comparator): Following a comprehensive evaluation,this group of subjects will undergo a 20-minute treatment once per week for four weeks.
  Interventions: Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology
- Non- DED Control Arm (Other): Following a comprehensive evaluation, this group of subjects will undergo a 20-minute treatment once per week for four weeks.
  Interventions: Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology
- DED Control Arm (Sham Comparator): Following a comprehensive evaluation, the sham treatment group will firstly undergo a 20-minute sham treatment once per week for four weeks. Two additional comprehensive evaluations and tear fluid collections will be conducted one month and three months after the completion of the treatment period. After the three-month post-treatment evaluation, the control group will receive four weekly treatments.
  Interventions: Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology

INTERVENTIONS:
Device: The Rexon-Eye, an electrotherapy device utilizing Quantum Molecular Resonance (QMR) technology — The device has received EC certification as a medical device for the treatment of ocular surface disorders. It will deliver a low-intensity alternating electrical current (ranging from 4 MHz to 64 MHz) to targeted biological tissue via contact electrodes. Previous studies have shown the effectiveness of this treatment in alleviating dry eye symptoms, both subjectively and objectively.

SUMMARY:
In this study, the initial tear proteome profiles in Dry Eye Disease (DED) patients, the safety and effectiveness of using an EC certificate DED treatment device in DED management, together with the associated global tear proteome changes, will be investigated.

DETAILED DESCRIPTION:
Diagnosis of Dry Eye Disease (DED) is current based on questionnaires, quantitative and qualitive tear and ocular surface assessment such as tear breakup time, corneal staining, and tear osmolarity. However, many of these clinical procedures show weak correlation between the clinical findings and subjective symptoms. Therefore, a more reliable method to aid in the diagnosis and management of dry eye disease is clearly needed.

Recently, a high frequency electrotherapy device using Quantum Molecular Resonance (QMR) technique, the Rexon-Eye was approved with EC certificate as a medical device for the treatment of the ocular surface disorders. During the treatment, a low-intensity, high-frequency (a spectrum of frequencies ranging from 4 MHz to 64 MHz) stimulations are applied on the epidermis of closed eyelids up to the lid border by special designed goggles. Previous data showed that it could effectively improve symptoms and clinical signs of DED by increasing the tear secretion and improving the meibomian gland function. Although clinically safe and effective, the mechanisms on how the stimulation could benefit DED are still unknown and ocular changes in response to the DED treatment in molecular level has not yet been investigated.

In this study, the initial tear proteome profiles in DED patients, the safety and effectiveness of using QMR in DED management together with the associated global tear proteome changes will be investigated. A total of 75 participants aged 18 to 65 years old will be recruited. 50 patients are DED patients and will be randomly assigned into treatment group and blinded control group. 25 non-DED age-matched subjects will be recruited as normal control. After the baseline DED evaluation, those eligible patients will be randomly allocated into treatment group and blinded control group. A total of four treatments will be performed to the treatment group and normal control in a weekly bases according the suggested protocol by the manufacturer. The blinded control group will receive sham treatments also in a weekly bases. Two outcome evaluation visits will be arranged for all participants one month and three months after the final treatment (i.e. the 4th treatment). The blinded control group will receive four QMR treatment after the second outcome evaluation visit. The same four treatments (identical to the treatment group) will be conducted followed by two extra outcome evaluation visits. Baseline and post-treatment tears will be collected using Schirmer strips, and changes in the tear proteome will be quantified using a mass spectrometer.

ELIGIBILITY:
Inclusion Criteria:

* OSDI score ≥ 13, and
* Fail one of the three diagnostic tests:

  * Non-invasive tear break-up time (NITBUT) less than 10s;
  * Tears osmolarity higher than or equals to 308 mOsm/L or inter-ocular difference > 8 mOsm/L;
  * When assessing with slit lamp, shows more than 9 spots of conjunctival stain with lissamine green, more than 5 spots of corneal stain with fluorescein or lid wiper epitheliopathy (LWE) with lissamine green ≥ 2 mm in length and/or ≥ 25% sagittal width.

Exclusion Criteria:

* Any active ocular infections, inflammations or anomalies in eyelid;
* Pregnant or lactating;
* Uncontrolled, newly diagnosed systemic diseases or with modified long-term medications within 6 months;
* Carrying active implantable devices (e.g., pacemakers and hearing aids)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical efficacy | From enrollment to the end of treatment at 4 (Treatment group) to 8 (Sham treatment group)months
  Ocular Surface Disease Index

SECONDARY OUTCOMES:
The associated tear proteomics changes after treatment | From enrollment to the end of treatment at 4 (Treatment group) to 8 (Sham treatment group)months
  Differences in tear protein groups induced by the treatment, along with their corresponding flow change relative to baseline will be investigated through mass spectrometry analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hei Jimmy Tse, Principal Investigator — The Hong Kong Polytechnic University, Hong Kong,
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong,, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trivli A, Karmiris E, Dalianis G, Ruggeri A, Terzidou C. Evaluating the efficacy of Quantum Molecular Resonance (QMR) electrotherapy in mixed-type dry eye patients. J Optom. 2023 Apr-Jun;16(2):128-134. doi: 10.1016/j.optom.2022.06.003. Epub 2022 Jul 16. PMID 35851496